CLINICAL TRIAL: NCT04812535
Title: Open Label, Multicenter Phase II Study of the C5a Antibody IFX-1 Alone or IFX-1 + Pembrolizumab in Patients With PD-1 or PD-L1 Resistant/Refractory Locally Advanced or Metastatic Cutaneous Squamous Cell Carcinoma (cSCC)
Brief Title: Non-comparative Study of IFX-1 Alone or IFX-1+Pembrolizumab in Patients With Locally Advanced or Metastatic cSCC.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decided to stop the development of vilobelimab in cSCC and early terminated the IFX-1-P2.8 trial due to new alternative treatments for cSCC with high efficacy rates.
Sponsor: InflaRx GmbH (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IFX-1 P2.8; MK-3475-A93 (Other: Merck Sharp & Dohme LLC); KEYNOTE-A93 (Other: Merck Sharp & Dohme LLC); 2020-000864-42 (EudraCT Number)
Record Dates: First submitted 2021-03-10; First posted 2021-03-23 (Actual); Results first posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: SCC - Squamous Cell Carcinoma of Skin
Keywords: cSCC; metastatic; locally advanced
MeSH Terms: conditions — Neoplasm Metastasis | interventions — vilobelimab; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Arm A: Vilobelimab monotherapy; Arm B: Vilobelimab + in combination with approved dosing scheme of pembrolizumab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A: (Experimental): Vilobelimab monotherapy; Vilobelimab monotherapy was administered as a 30-minute (-5 / +10 minutes) intravenous infusion as follows: 800 mg on Days 1, 4, 8, and 15, followed by 1600 mg Q2W starting on Day 22 of Cycle 1 until end of treatment (EOT)
  Interventions: Drug: Vilobelimab
- Arm B: Regimen 1: (Experimental): Vilobelimab + pembrolizumab combination therapy; Vilobelimab was administered as a 30-minute (-5/+10 minutes) intravenous infusion as follows: 400 mg on Days 1, 4, 8, and 15, followed by 800 mg Q2W starting on Day 22 of Cycle 1 until EOT. Vilobelimab treatment was combined with pembrolizumab, administered as a 30-minute (-5/+10 minutes) intravenous infusion at a dose of 400 mg starting at Day 8 of Cycle 1 and then Q6W on Day 1 of each treatment cycle
  Interventions: Drug: Vilobelimab + pembrolizumab combination therapy
- Arm B: Regimen 2: (Experimental): Vilobelimab + pembrolizumab combination therapy; Vilobelimab was administered as a 30-minute (-5/+10 minutes) intravenous infusion as follows: 600 mg on Days 1, 4, 8, and 15, followed by 1200 mg Q2W starting on Day 22 of Cycle 1 until EOT. Vilobelimab treatment was combined with pembrolizumab, administered as a 30-minute (-5/+10 minutes) intravenous infusion at a dose of 400 mg starting at Day 8 of Cycle 1 and then Q6W on Day 1 of each treatment cycle
  Interventions: Drug: Vilobelimab + pembrolizumab combination therapy
- Arm B: Regimen 3: (Experimental): Vilobelimab + pembrolizumab combination therapy; Vilobelimab was administered as a 30-minute (-5/+10 minutes) intravenous infusion as follows: 800 mg on Days 1, 4, 8, and 15, followed by 1600 mg Q2W starting on Day 22 of Cycle 1 until EOT. Vilobelimab treatment was combined with pembrolizumab, administered as a 30-minute (-5/+10 minutes) intravenous infusion at a dose of 400 mg starting at Day 8 of Cycle 1 and then Q6W on Day 1 of each treatment cycle
  Interventions: Drug: Vilobelimab + pembrolizumab combination therapy

INTERVENTIONS:
Drug: Vilobelimab — Vilobelimab Monotherapy
  Arms: Arm A:
Drug: Vilobelimab + pembrolizumab combination therapy — Vilobelimab + pembrolizumab combination therapy
  Other Names: KEYTRUDA®
  Arms: Arm B: Regimen 1:; Arm B: Regimen 2:; Arm B: Regimen 3:

SUMMARY:
This is an open-label, "non comparative", non-randomized, Phase II study. Patients will be enrolled in 2 treatment arms

DETAILED DESCRIPTION:
This is an open-label, non-randomized, Phase II study. Patients will be enrolled in 2 treatment arms (Arm A: Vilobelimab monotherapy; Arm B: Vilobelimab + pembrolizumab combination therapy), both consisting of 2 stages whereas Arm B starts with a safety run in portion. Enrollment follows an optimal Simon's 2-stage design with an interim analysis of treatment response after Stage 1 prior to patient enrollment into Stage 2.

Arm B will start after ≥3 patients have been treated in Arm A and no toxicity concerns have emerged. In a safety run-in part of Arm B, escalating doses of Vilobelimab will be investigated in combination with pembrolizumab in order to identify the maximum tolerated dose (MTD) or recommended Phase II dose (RP2D). Patients will be treated until progression, occurrence of unacceptable toxicity, or treatment discontinuation for any other reason.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age on day of signing informed consent
* Patients with biopsy-proven, histologically or cytologically confirmed (a.) locally advanced cSCC not amenable for curative treatment or (b.) metastatic cSCC. Patients must have been treated with all approved therapies for (a.) inoperable locally advanced cSCC contraindicated for radiation therapy or (b.) metastatic cSCC. All patients to be included must have progressed on PD-1- or PD-L1-inhibitory antibody therapy.
* Patients must have progressed on treatment with an anti-PD-1/L1 monoclonal antibody (mAb) administered either as monotherapy or in combination with other checkpoint inhibitors or other therapies. PD-1 treatment progression is defined by meeting all of the following criteria:

  1. Has received ≥2 doses of an anti-PD-1/L1 mAb that has been approved for treatment of cSCC or any solid tumor
  2. Has demonstrated PD/iCPD after PD-1/L1 inhibitor treatment as defined by RECIST v1.1/iRECIST. The initial evidence of disease progression is to be confirmed by a second assessment ≥4 weeks from the date of the first documented disease progression, unless there is rapid clinical progression.
  3. Disease progression has been documented within 12 weeks from the last dose of anti-PD-1/L1 mAb.
* The PD-1-/PD-L1 infusion must have been the most recent treatment for locally advanced or metastatic cSCC.
* In addition to providing the material for ensuring the diagnosis as stated in inclusion criterion 2a for patients with locally advanced cSCC, patients must consent to undergo the following biopsies (at each time point a punch biopsy of externally visible cSCC lesions or a biopsy of material from accessible metastases) for biomarker assessments:

  1. At baseline prior to the first administration of the investigational therapy and if possible, within 7 days prior to initiation of study treatment administration (mandatory for all patients)
  2. For Stage 2 patients only: on Cycle 2 Day 1 (±3 days) (mandatory)
  3. For Stage 2 patients only: at the time of CR/iCR/PR/iPR (optional, to be conducted only if the investigator considers this biopsy as clinically possible and potentially informative)
  4. For Stage 2 patients only: At the time of tumor progression (optional, to be conducted only if the investigator considers this biopsy as clinically possible and potentially informative).
* Patients must have the following minimum washout before first study treatment administration from previous treatments:

  1. ≥4 weeks for mAbs, systemic cytotoxic anticancer therapy, treatment with other anticancer investigational agents
  2. ≥3 weeks for local radiation therapy
* Eastern Cooperative Oncology Group performance status (ECOG PS) status of ≤1
* Adequate organ function
* Patient (or legally acceptable representative if applicable) provides written informed consent for the study.

Exclusion Criteria:

* Patients with limited cSCC, who do not require systemic therapy
* Has known active central nervous system metastases and/or carcinomatous meningitis.

Patients with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for ≥4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for ≥14 days prior to first dose of study treatment.

* Has a diagnosis of immunodeficiency or autoimmune disease, or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 3 weeks prior the first dose of study treatment
* Patients who have a history of (non-infectious) pneumonitis that required steroids or have current pneumonitis
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent, or with an agent directed to another stimulatory or co-inhibitory T cell receptor (e.g., cytotoxic T-lymphocyte-associated antigen 4, OX 40, CD137) and was discontinued from that treatment due to a ≥Grade 3 irAE
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab or IFX-1 and/or any of their excipients or had a severe (≥Grade 3) infusion-related reaction to treatments with other mAbs
* Patients who fulfil inclusion criterion 6 (washout times) but who have not recovered from side effects of such therapies
* Has received a live vaccine within 30 days prior to the first dose of study treatment
* Patients who have undergone major surgery <4 weeks prior to starting study treatment
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment
* Patients with known ≥Grade 3 (per National Cancer Institute common terminology criteria for adverse events [NCI CTCAE] v5.0 criteria) active systemic or cutaneous viral, bacterial, or fungal infection
* Patients with known history of Hepatitis B or C infections or known to be positive for Hepatitis B antigen (HBsAg)/ Hepatitis B virus (HBV) DNA or Hepatitis C Antibody or RNA. Active Hepatitis C is defined by a known positive Hep C Ab result and known quantitative HCV RNA results greater than the lower limits of detection of the assay.
* Patients who have a history of human immunodeficiency virus infection
* Patients who have a history of interstitial lung disease
* Patients who have had an allogeneic tissue/solid organ transplant
* Patients with a history of other malignancies during the past 5 years.
* Patients who are pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 3 months after the last dose of IFX-1 or 120 days after the last dose of pembrolizumab
* Women of childbearing potential (WOCBP) who have a positive serum pregnancy test result within 7 days before treatment
* Male patients and WOCBP who do not agree to practice an effective method of contraception during study and until 3 months after last dose of IFX-1 or 120 days after last dose of pembrolizumab
* Patients with congestive heart failure, Class III or IV, by New York Heart Association criteria
* Patients with any serious underlying medical condition that would impair their ability to receive or tolerate the planned treatment
* Patients with dementia or altered mental status that would preclude understanding and rendering of informed consent document

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. D. Schadendorf, MD, Principal Investigator — University Hospital, Essen
Locations (25):
- United States (6):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Anschutz Cancer Pavilion, Aurora, Colorado
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Orlando Health, Inc., Orlando, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Inova Schar Cancer Institute, Fairfax, Virginia
- Belgium (2):
  - University Hospital Antwerp (UZA), Edegem
  - St. Augustinus Hospital, Wilrijk
- France (5):
  - University Hospital Center of Grenoble Alpes, Department of Dermatology, Grenoble
  - South Lyon Hospital Center, Lyon
  - CHU APHM la Timone / Aix Marseille University, Dermatology and Skin Cancer Department, Marseille
  - St. Louis Hospital, Paris
  - University Hospital Center of Poitiers, Department of Oncology, Poitiers
- Germany (7):
  - University Hospital Erlangen, Department of Dermatology, Erlangen
  - University Duisburg-Essen, University Hospital Essen, Department of Dermatology, Essen
  - Frankfurt University Clinic, Department of Dermatology, Venereology and Allergology, Frankfurt
  - University Hospital Hamburg-Eppendorf, Hamburg
  - University Hospital Leipzig, Department of Dermatology, Venereology and Allergology, Leipzig
  - University Hospital Regensburg, Clinic and Policlinic for Dermatology, Regensburg
  - University Hospital Tuebingen, Department of Dermatology, Tübingen
- Spain (5):
  - University Hospital Vall d'Hebron, Barcelona
  - ICO Hospitalet, Barcelona
  - MD Anderson International Cancer Center Spain, Madrid
  - Regional University Hospital of Malaga, Málaga
  - University Clinical Hospital of Salamanca, Salamanca

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: According to protocol stipulations, a participant is enrolled into the study if informed consent form is completed (signed and dated). This reflects the "Protocol Enrollment: 30" participant number. Five (5) participants failed screening (after ICF signed) and were not assigned to and treated in the different Arms/Groups, constituting the "Total Started in Participant Flow: 25" participant number.
Groups:
- Arm A:: Vilobelimab monotherapy; Vilobelimab monotherapy was administered as a 30-minute (-5 / +10 minutes) intravenous infusion as follows: 800 mg on Days 1, 4, 8, and 15, followed by 1600 mg Q2W starting on Day 22 of Cycle 1 until EOT
Period: Overall Study
Arm/Group | Arm A: | Arm B: Regimen 1: | Arm B: Regimen 2: | Arm B: Regimen 3:
Started | 10 | 3 | 6 | 6
Completed | 1 | 1 | 1 | 1
Not Completed | 9 | 2 | 5 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Death | 7 | 2 | 4 | 1
Not completed — Due to premature study termination by sponsor | 2 | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: | Arm B: Regimen 1: | Arm B: Regimen 2: | Arm B: Regimen 3: | Total
Number analyzed (Participants) | 10 | 3 | 6 | 6 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.0 (13.4) | 81.3 (13.3) | 72.8 (10.6) | 70.8 (9.6) | 73.8 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 4 | 5 | 16
  Male | 5 | 1 | 2 | 1 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 10 | 3 | 5 | 6 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 9 | 3 | 6 | 6 | 24
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 0 | 2 | 1 | 0 | 3
  United States | 1 | 0 | 0 | 2 | 3
  France | 3 | 1 | 0 | 0 | 4
  Germany | 5 | 0 | 3 | 2 | 10
  Spain | 1 | 0 | 2 | 2 | 5
Weight at screening [Mean (Standard Deviation); unit: kilogram] | 82.56 (45.40) | 73.33 (21.57) | 71.12 (16.44) | 71.48 (9.59) | 76.05 (30.29)
Height at screening [Mean (Standard Deviation); unit: centimeter] | 167.7 (12.1) | 167.0 (2.6) | 160.3 (5.9) | 169.0 (9.8) | 166.2 (9.7)
BMI at screening [Mean (Standard Deviation); unit: kg/m²] | 29.08 (14.18) | 26.13 (6.79) | 27.90 (7.22) | 25.10 (3.48) | 27.49 (9.76)
Duration of cSCC [Mean (Standard Deviation); unit: years] | 4.4 (7.4) | 5.0 (1.0) | 3.3 (2.1) | 4.0 (3.5) | 4.1 (4.9)
Primary diagnosis [Count of Participants; unit: Participants]
  Locally advanced cSCC | 6 | 1 | 1 | 2 | 10
  Metastatic cSCC | 4 | 2 | 5 | 4 | 15
Tumor category (TNM staging at initial diagnosis) [Count of Participants; unit: Participants] — Primary diagnosis: Metastatic cSCC was considered worse outcome as compared to Locally advanced cSCC according to NCCN Guidelines Squamous Cell Skin Cancer V1.2024 (latest version) and AJCC TNM Staging Classification, 8th Ed., 2017. Tumor category (TNM staging at initial diagnosis): ascending T categories from TX to T4 were considered increasing worse outcome according to NCCN Guidelines Squamous Cell Skin Cancer V1.2024 (latest version) and AJCC TNM Staging Classification, 8th Ed., 2017.
  Participants
    TX | 1 | 0 | 0 | 1 | 2
    Tis | 0 | 0 | 0 | 0 | 0
    T1 | 1 | 2 | 3 | 2 | 8
    T2 | 2 | 0 | 1 | 0 | 3
    T3 | 4 | 1 | 0 | 1 | 6
    T4 | 2 | 0 | 2 | 2 | 6
Nodes (TNM staging at initial diagnosis) [Count of Participants; unit: Participants] — Nodes (TNM staging at initial diagnosis): ascending N categories from NX to N3 were considered increasing worse outcome according to NCCN Guidelines Squamous Cell Skin Cancer V1.2024 (latest version) and AJCC TNM Staging Classification, 8th Ed., 2017.
  Participants
    NX | 2 | 1 | 1 | 0 | 4
    N0 | 6 | 2 | 2 | 4 | 14
    N1 | 1 | 0 | 1 | 0 | 2
    N2 | 0 | 0 | 2 | 0 | 2
    N3 | 1 | 0 | 0 | 2 | 3
Metastases (TNM staging at initial diagnosis) [Count of Participants; unit: Participants] — Metastasis (TNM staging at initial diagnosis): ascending M categories from M0 to M1 were considered increasing worse outcome according to NCCN Guidelines Squamous Cell Skin Cancer V1.2024 (latest version) and AJCC TNM Staging Classification, 8th Ed., 2017.
  Participants
    M0 | 10 | 3 | 5 | 5 | 23
    M1 | 0 | 0 | 1 | 1 | 2
Histologic grade (TNM staging at initial diagnosis) [Count of Participants; unit: Participants] — Histologic grade (TNM staging at initial diagnosis): ascending G categories from GX to G4 were considered increasing worse outcome according to NCCN Guidelines Squamous Cell Skin Cancer V1.2024 (latest version) and AJCC TNM Staging Classification, 8th Ed., 2017.
  Participants
    GX | 1 | 1 | 1 | 1 | 4
    G1 | 3 | 0 | 0 | 2 | 5
    G2 | 2 | 2 | 2 | 2 | 8
    G3 | 2 | 0 | 3 | 0 | 5
    G4 | 0 | 0 | 0 | 0 | 0
    Missing | 2 | 0 | 0 | 1 | 3
Prognostic stage group [Count of Participants; unit: Participants] — Prognostic stage group table, comparing TNM staging at initial diagnosis versus TNM staging at study entry: ascending stage categories from Stage 0 to Stage IV were considered increasing worse outcome according to NCCN Guidelines Squamous Cell Skin Cancer V1.2024 (latest version) and AJCC TNM Staging Classification, 8th Ed., 2017.
  Participants
    TNM staging at initial diagnosis: Stage 0 | 0 | 0 | 0 | 0 | 0
    TNM staging at initial diagnosis: Stage I | 1 | 2 | 1 | 2 | 6
    TNM staging at initial diagnosis: Stage II | 2 | 0 | 1 | 0 | 3
    TNM staging at initial diagnosis: Stage III | 3 | 1 | 1 | 1 | 6
    TNM staging at initial diagnosis: Stage IV | 3 | 0 | 3 | 2 | 8
    TNM staging at initial diagnosis: Missing | 1 | 0 | 0 | 1 | 2
    TNM staging at study entry: Stage 0 | 0 | 0 | 0 | 0 | 0
    TNM staging at study entry: Stage I | 0 | 0 | 0 | 0 | 0
    TNM staging at study entry: Stage II | 0 | 0 | 0 | 0 | 0
    TNM staging at study entry: Stage III | 2 | 0 | 0 | 1 | 3
    TNM staging at study entry: Stage IV | 8 | 3 | 6 | 5 | 22
    TNM staging at study entry: Missing | 0 | 0 | 0 | 0 | 0
Prognostic staging system [Count of Participants; unit: Participants] — Prognostic staging system table: 4 prognostic staging systems (AJCC8, AJCC 7, BHW, Other) according to which cSCC TNM staging at initial diagnosis versus TNM staging at study entry were performed.
  Participants
    TNM staging at initial diagnosis: AJCC 8 | 5 | 3 | 6 | 5 | 19
    TNM staging at initial diagnosis: AJCC 7 | 3 | 0 | 0 | 0 | 3
    TNM staging at initial diagnosis: BHW | 0 | 0 | 0 | 0 | 0
    TNM staging at initial diagnosis: Other | 1 | 0 | 0 | 0 | 1
    TNM staging at initial diagnosis: Missing | 1 | 0 | 0 | 1 | 2
    TNM staging at study entry: AJCC 8 | 6 | 3 | 6 | 5 | 20
    TNM staging at study entry: AJCC 7 | 3 | 0 | 0 | 0 | 3
    TNM staging at study entry: BHW | 0 | 0 | 0 | 0 | 0
    TNM staging at study entry: Other | 1 | 0 | 0 | 1 | 2
    TNM staging at study entry: Missing | 0 | 0 | 0 | 0 | 0
H&P Location/size - area L [Count of Participants; unit: Participants] — H&P Location/size - area L table: Split into risk groups according to disease history and physical parameters (H&P) Location/size for area L (low risk: trunk, extremities) defined by < 20 mm and >= 20 mm according to NCCN Guidelines Squamous Cell Skin Cancer V1.2024 (latest version).
  Participants
    <20 mm | 1 | 1 | 2 | 1 | 5
    >=20 mm | 3 | 1 | 2 | 1 | 7
    Missing | 6 | 1 | 2 | 4 | 13
H&P Location/size - area M [Count of Participants; unit: Participants] — H&P Location/size - area M table: Split into risk groups according to disease history and physical parameters (H&P) Location/size for area M (medium risk: cheeks, forehead, neck, scalp) defined by < 10 mm and >= 10 mm according to NCCN Guidelines Squamous Cell Skin Cancer V1.2024 (latest version).
  Participants
    <10 mm | 1 | 1 | 0 | 0 | 2
    >=10 mm | 5 | 1 | 3 | 3 | 12
    Missing | 4 | 1 | 3 | 3 | 11
H&P Location/size - area H [Count of Participants; unit: Participants] — H&P Location/size - area H table: Split into risk groups according to disease history and physical parameters (H&P) Location/size for area H (high risk: face, ears, genitals, hands, feet) defined by 'No' and 'Yes' according to NCCN Guidelines Squamous Cell Skin Cancer V1.2024 (latest version).
  Participants
    No | 4 | 0 | 2 | 0 | 6
    Yes | 4 | 3 | 1 | 2 | 10
    Missing | 2 | 0 | 3 | 4 | 9
H&P Borders [Count of Participants; unit: Participants] — H&P Borders table: Split into risk groups according to cSCC lesion borders defined by 'Well defined' (low risk) and 'Poorly defined' (high risk) according to NCCN Guidelines Squamous Cell Skin Cancer V1.2024 (latest version).
  Participants
    Well defined | 4 | 2 | 3 | 2 | 11
    Poorly defined | 4 | 1 | 1 | 1 | 7
    Missing | 2 | 0 | 2 | 3 | 7
H&P Primary vs recurrent [Count of Participants; unit: Participants] — H&P Primary vs recurrent table: Split into risk groups according to primary versus recurrent cSCC disease defined by 'Primary' (low risk) and 'Recurrent' (high risk) according to NCCN Guidelines Squamous Cell Skin Cancer V1.2024 (latest version).
  Participants
    Primary | 3 | 0 | 3 | 3 | 9
    Recurrent | 7 | 3 | 3 | 1 | 14
    Missing | 0 | 0 | 0 | 2 | 2
H&P Immunosuppression [Count of Participants; unit: Participants]
  - | 10 | 3 | 6 | 4 | 23
  + | 0 | 0 | 0 | 1 | 1
  Missing | 0 | 0 | 0 | 1 | 1
H&P Site of prior RT or chronic inflammatory process [Count of Participants; unit: Participants]
  - | 6 | 2 | 4 | 3 | 15
  + | 4 | 1 | 2 | 1 | 8
  Missing | 0 | 0 | 0 | 2 | 2
H&P Rapidly growing tumour [Count of Participants; unit: Participants]
  - | 4 | 1 | 4 | 3 | 12
  + | 6 | 2 | 2 | 1 | 11
  Missing | 0 | 0 | 0 | 2 | 2
H&P Neurologic symptoms [Count of Participants; unit: Participants]
  - | 9 | 3 | 6 | 5 | 23
  + | 1 | 0 | 0 | 0 | 1
  Missing | 0 | 0 | 0 | 1 | 1
Pathology Degree of differentiation [Count of Participants; unit: Participants]
  Well or moderately differentiated | 7 | 2 | 2 | 5 | 16
  Poorly differentiated | 3 | 1 | 4 | 0 | 8
  Missing | 0 | 0 | 0 | 1 | 1
Pathology Acantholytic, adenosquamous, desmoplastic, or metaplastic subtypes [Count of Participants; unit: Participants]
  - | 9 | 2 | 5 | 3 | 19
  + | 0 | 1 | 0 | 1 | 2
  Missing | 1 | 0 | 1 | 2 | 4
Pathology Depth: thickness or level of invasion [Count of Participants; unit: Participants]
  <=6 mm and no invasion beyond subcutaneous fat | 3 | 2 | 2 | 2 | 9
  >6 mm or invasion beyond subcutaneous fat | 6 | 1 | 2 | 2 | 11
  Missing | 1 | 0 | 2 | 2 | 5
Pathology Perineural, lymphatic or vascular involvement [Count of Participants; unit: Participants]
  - | 5 | 1 | 3 | 3 | 12
  + | 4 | 2 | 1 | 1 | 8
  Missing | 1 | 0 | 2 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response Rate (Best ORR) - Arm A and Arm B
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) and immunologic RECIST (iRECIST) for target lesions and assessed by computed tomography (CT) or magnetic resonance imaging (MRI). Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): ≥30% decrease in the sum of the diameters of target lesions; Best Overall Response (OR) = CR + PR, from the start of the treatment until PD/recurrence.
Time Frame: Up to 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: | Arm B: Regimen 1: | Arm B: Regimen 2: | Arm B: Regimen 3:
Number analyzed (Participants) | 10 | 3 | 6 | 6
Participants
  ORR (Responder) | 1 | 0 | 1 | 2
  Non-responder | 9 | 3 | 4 | 4
  No post baseline measurement | 0 | 0 | 1 | 0

2. Primary Outcome: Dose-limiting Toxicity (DLT) - Arm B
Description: Frequency of dose-limiting toxicities (DLTs) by dose cohort.
Time Frame: Cycle 1 Day 1 - Cycle 1 Day 36
Measure: Count of Participants; unit: Participants
Groups:
- Arm B Regimen 1:: Vilobelimab + pembrolizumab combination therapy; Vilobelimab was administered as a 30-minute (-5/+10 minutes) intravenous infusion as follows: 400 mg on Days 1, 4, 8, and 15, followed by 800 mg Q2W starting on Day 22 of Cycle 1 until EOT. Vilobelimab treatment was combined with pembrolizumab, administered as a 30-minute (-5/+10 minutes) intravenous infusion at a dose of 400 mg starting at Day 8 of Cycle 1 and then Q6W on Day 1 of each treatment cycle
- Arm B Regimen 2:: Vilobelimab + pembrolizumab combination therapy; Vilobelimab was administered as a 30-minute (-5/+10 minutes) intravenous infusion as follows: 600 mg on Days 1, 4, 8, and 15, followed by 1200 mg Q2W starting on Day 22 of Cycle 1 until EOT. Vilobelimab treatment was combined with pembrolizumab, administered as a 30-minute (-5/+10 minutes) intravenous infusion at a dose of 400 mg starting at Day 8 of Cycle 1 and then Q6W on Day 1 of each treatment cycle
- Arm B Regimen 3:: Vilobelimab + pembrolizumab combination therapy; Vilobelimab was administered as a 30-minute (-5/+10 minutes) intravenous infusion as follows: 800 mg on Days 1, 4, 8, and 15, followed by 1600 mg Q2W starting on Day 22 of Cycle 1 until EOT.
  Vilobelimab treatment was combined with pembrolizumab, administered as a 30-minute (-5/+10 minutes) intravenous infusion at a dose of 400 mg starting at Day 8 of Cycle 1 and then Q6W on Day 1 of each treatment cycle
Arm/Group | Arm A: | Arm B Regimen 1: | Arm B Regimen 2: | Arm B Regimen 3:
Number analyzed (Participants) | 10 | 3 | 6 | 6
Participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Disease Control Rate - Arm A and Arm B
Description: Disease control rate is defined as the relative number of patients achieving stable disease (SD/iSD), CR/iCR or PR/iPR according to modified RECIST v1.1 (including clinical response)/iRECIST response.
Time Frame: Up to 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: | Arm B: Regimen 1: | Arm B: Regimen 2: | Arm B: Regimen 3:
Number analyzed (Participants) | 10 | 3 | 6 | 6
Participants
  Cycle 2 Day 1: Controlled disease | 2 | 0 | 3 | 4
  Cycle 2 Day 1: No controlled disease | 6 | 1 | 2 | 2
  Cycle 2 Day 1: No response assessment | 2 | 2 | 1 | 0
  Cycle 3 Day 1: Controlled disease | 1 | 0 | 1 | 2
  Cycle 3 Day 1: No controlled disease | 0 | 0 | 1 | 2
  Cycle 3 Day 1: No response assessment | 9 | 3 | 4 | 2
  Cycle 3 Day 29: Controlled disease | 1 | 0 | 0 | 0
  Cycle 3 Day 29: No controlled disease | 0 | 0 | 0 | 0
  Cycle 3 Day 29: No response assessment | 9 | 3 | 6 | 6
  Cycle 4 Day 1: Controlled disease | 1 | 0 | 1 | 2
  Cycle 4 Day 1: No controlled disease | 0 | 0 | 0 | 1
  Cycle 4 Day 1: No response assessment | 9 | 3 | 5 | 3
  Cycle 5 Day 1: Controlled disease | 2 | 0 | 1 | 2
  Cycle 5 Day 1: No controlled disease | 0 | 0 | 0 | 0
  Cycle 5 Day 1: No response assessment | 8 | 3 | 5 | 4
  Cycle 6 Day 1: Controlled disease | 2 | 0 | 1 | 2
  Cycle 6 Day 1: No controlled disease | 0 | 0 | 0 | 0
  Cycle 6 Day 1: No response assessment | 8 | 3 | 5 | 4
  Cycle 7 Day 1: Controlled disease | 2 | 0 | 1 | 1
  Cycle 7 Day 1: No controlled disease | 0 | 0 | 0 | 0
  Cycle 7 Day 1: No response assessment | 8 | 3 | 5 | 5
  Cycle 8 Day 1: Controlled disease | 1 | 0 | 1 | 0
  Cycle 8 Day 1: No controlled disease | 0 | 0 | 0 | 1
  Cycle 8 Day 1: No response assessment | 9 | 3 | 5 | 5
  Cycle 9 Day 1: Controlled disease | 2 | 0 | 1 | 0
  Cycle 9 Day 1: No controlled disease | 0 | 0 | 0 | 0
  Cycle 9 Day 1: No response assessment | 8 | 3 | 5 | 6
  Cycle 10 Day 1: Controlled disease | 1 | 0 | 1 | 0
  Cycle 10 Day 1: No controlled disease | 0 | 0 | 0 | 0
  Cycle 10 Day 1: No response assessment | 9 | 3 | 5 | 6
  Cycle 11 Day 1: Controlled disease | 2 | 0 | 1 | 0
  Cycle 11 Day 1: No controlled disease | 0 | 0 | 0 | 0
  Cycle 11 Day 1: No response assessment | 8 | 3 | 5 | 6
  Cycle 12 Day 1: Controlled disease | 0 | 0 | 1 | 0
  Cycle 12 Day 1: No controlled disease | 0 | 0 | 0 | 0
  Cycle 12 Day 1: No response assessment | 10 | 3 | 5 | 6
  Cycle 12 Day 29: Controlled disease | 1 | 0 | 0 | 0
  Cycle 12 Day 29: No controlled disease | 0 | 0 | 0 | 0
  Cycle 12 Day 29: No response assessment | 9 | 3 | 6 | 6
  Cycle 13 Day 1: Controlled disease | 0 | 0 | 1 | 0
  Cycle 13 Day 1: No controlled disease | 1 | 0 | 0 | 0
  Cycle 13 Day 1: No response assessment | 9 | 3 | 5 | 6
  Cycle 14 Day 1: Controlled disease | 0 | 0 | 1 | 0
  Cycle 14 Day 1: No controlled disease | 0 | 0 | 0 | 0
  Cycle 14 Day 1: No response assessment | 10 | 3 | 5 | 6
  Cycle 14 Day 15: Controlled disease | 0 | 0 | 0 | 0
  Cycle 14 Day 15: No controlled disease | 1 | 0 | 0 | 0
  Cycle 14 Day 15: No response assessment | 9 | 3 | 6 | 6
  Cycle 15 Day 1: Controlled disease | 0 | 0 | 1 | 0
  Cycle 15 Day 1: No controlled disease | 1 | 0 | 0 | 0
  Cycle 15 Day 1: No response assessment | 9 | 3 | 5 | 6
  Cycle 16 Day 1: Controlled disease | 0 | 0 | 1 | 0
  Cycle 16 Day 1: No controlled disease | 0 | 0 | 0 | 0
  Cycle 16 Day 1: No response assessment | 10 | 3 | 5 | 6
  Cycle 17 Day 1: Controlled disease | 0 | 0 | 1 | 0
  Cycle 17 Day 1: No controlled disease | 0 | 0 | 0 | 0
  Cycle 17 Day 1: No response assessment | 10 | 3 | 5 | 6
  EOT Visit: Controlled disease | 0 | 0 | 1 | 0
  EOT Visit: No controlled disease | 3 | 2 | 0 | 3
  EOT Visit: No response assessment | 7 | 1 | 5 | 3

4. Secondary Outcome: Progression-free Survival (PFS)- Arm A and Arm B
Description: PFS is defined as the time from first study treatment administration to progression (i.e. PD, iUPD, iCPD) or death. Patients without progression are censored at their last visit/study treatment administration.
Time Frame: Up to 36 months
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Arm A:: Vilobelimab monotherapy Vilobelimab monotherapy was administered as a 30-minute (-5 / +10 minutes) intravenous infusion as follows: 800 mg on Days 1, 4, 8, and 15, followed by 1600 mg Q2W starting on Day 22 of Cycle 1 until EOT
- Arm B Regimen 1:: Vilobelimab + pembrolizumab combination therapy Vilobelimab was administered as a 30-minute (-5/+10 minutes) intravenous infusion as follows: 400 mg on Days 1, 4, 8, and 15, followed by 800 mg Q2W starting on Day 22 of Cycle 1 until EOT. Vilobelimab treatment was combined with pembrolizumab, administered as a 30-minute (-5/+10 minutes) intravenous infusion at a dose of 400 mg starting at Day 8 of Cycle 1 and then Q6W on Day 1 of each treatment cycle
- Arm B Regimen 2:: Vilobelimab + pembrolizumab combination therapy Vilobelimab was administered as a 30-minute (-5/+10 minutes) intravenous infusion as follows: 600 mg on Days 1, 4, 8, and 15, followed by 1200 mg Q2W starting on Day 22 of Cycle 1 until EOT. Vilobelimab treatment was combined with pembrolizumab, administered as a 30-minute (-5/+10 minutes) intravenous infusion at a dose of 400 mg starting at Day 8 of Cycle 1 and then Q6W on Day 1 of each treatment cycle
- Arm B Regimen 3:: Vilobelimab + pembrolizumab combination therapy Vilobelimab was administered as a 30-minute (-5/+10 minutes) intravenous infusion as follows: 800 mg on Days 1, 4, 8, and 15, followed by 1600 mg Q2W starting on Day 22 of Cycle 1 until EOT. Vilobelimab treatment was combined with pembrolizumab, administered as a 30-minute (-5/+10 minutes) intravenous infusion at a dose of 400 mg starting at Day 8 of Cycle 1 and then Q6W on Day 1 of each treatment cycle
Arm/Group | Arm A: | Arm B Regimen 1: | Arm B Regimen 2: | Arm B Regimen 3:
Number analyzed (Participants) | 10 | 3 | 6 | 6
days | 50.0 [40.0 to 51.0] | 106.0 [43.0 to 106.0] | 90.0 [52.0 to NA] — The upper confidence limit is not calculable because the number of participants with event is insufficient | 87.5 [49.0 to NA] — The upper confidence limit is not calculable because the number of participants with event is insufficient

5. Secondary Outcome: Overall Survival (OS)- Arm A and Arm B
Description: Overall survival is defined as the time from first study treatment administration to death. Patients alive when they discontinue the study are censored at their last recorded date of being alive.
Time Frame: Up to 36 months
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Arm A: | Arm B: Regimen 1: | Arm B: Regimen 2: | Arm B: Regimen 3:
Number analyzed (Participants) | 10 | 3 | 6 | 6
days | 285.0 [52.0 to NA] — The upper confidence limit is not calculable because the number of participants with event is insufficient | 106.0 [63.0 to NA] — The upper confidence limit is not calculable because the number of participants with event is insufficient | 300.5 [103.0 to NA] — The upper confidence limit is not calculable because the number of participants with event is insufficient | NA [77.0 to NA] — The median and upper confidence limit is not calculable because the number of participants with event is insufficient

6. Secondary Outcome: Antidrug Antibodies (ADAs) - Arm A and Arm B
Description: Development of human antidrug antibodies (ADAs) against Vilobelimab. In contrast to the time frame of the secondary efficacy outcome measures (3.-5., 7.-8), which were reported until EOS (up to 36 months), the time frames of ADAs (6.) and PK (9.) are measured (only) until first FU. Therefore, the time frame is different, i.e. 24 months of treatment until EOT + (approx.) 12 weeks/3 months until first FU up to 27 months.
Time Frame: Up to 27 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: | Arm B Regimen 1: | Arm B Regimen 2: | Arm B Regimen 3:
Number analyzed (Participants) | 10 | 3 | 6 | 6
Participants
  Patients with at least one positive result | 2 | 0 | 0 | 0
  Patients without positive result | 8 | 3 | 6 | 6

7. Secondary Outcome: Quality of Life (QoL) - Arm A and Arm B
Description: The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-C30 version 3.0 measures the different aspects that define the quality of life of cancer patients or survivors. The reported total score ranges from 0 to 100 whereas a higher score represents a higher response level. The total score was calculated as mean of all 15 single scores. It was only calculated if all 15 single scores were non-missing (for more information see Fayers PM, Aaronson NK, Bjordal K, Groenvold M, Curran D, Bottomley A, on behalf of the EORTC Quality of Life Group. The EORTC QLQ-C30 Scoring Manual (3rd Edition). Published by: European Organisation for Research and Treatment of Cancer, Brussels 2001.). The absolute changes from baseline are presented.
Time Frame: Up to 36 months
Population: Not all patients are analyzed at each visit as the values for these patients are missing. This reason for this is either that the values for these patients are missing in the data or that these patients have already discontinued the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm A: | Arm B: Regimen 1: | Arm B: Regimen 2: | Arm B: Regimen 3:
Number analyzed (Participants) | 10 | 3 | 6 | 6
units on a scale
  Cycle 2 Day 1: number analyzed (Participants) | 7 | 1 | 4 | 5
  Cycle 2 Day 1 | 0.31 (4.38) | -0.80 (NA) — The standard deviation is not calculable, because the number of participants with available values at this visit and treatment group is one. | -2.68 (3.58) | -3.04 (6.21)
  Cycle 3 Day 1: number analyzed (Participants) | 2 | 0 | 2 | 3
  Cycle 3 Day 1 | -0.35 (5.73) |  | 3.00 (5.66) | -3.27 (1.62)
  Cycle 4 Day 1: number analyzed (Participants) | 2 | 0 | 1 | 2
  Cycle 4 Day 1 | 1.95 (0.21) |  | -2.40 (NA) — The standard deviation is not calculable, because the number of participants with available values at this visit and treatment group is one. | -6.35 (0.78)
  Cycle 5 Day 1: number analyzed (Participants) | 2 | 0 | 1 | 2
  Cycle 5 Day 1 | -1.15 (2.19) |  | -3.80 (NA) — The standard deviation is not calculable, because the number of participants with available values at this visit and treatment group is one. | -3.20 (2.83)
  Cycle 6 Day 1: number analyzed (Participants) | 2 | 0 | 1 | 2
  Cycle 6 Day 1 | 0.75 (0.49) |  | -1.40 (NA) — The standard deviation is not calculable, because the number of participants with available values at this visit and treatment group is one. | -1.85 (2.33)
  Cycle 7 Day 1: number analyzed (Participants) | 2 | 0 | 1 | 1
  Cycle 7 Day 1 | 2.55 (1.63) |  | 1.20 (NA) — The standard deviation is not calculable, because the number of participants with available values at this visit and treatment group is one. | -3.50 (NA) — The standard deviation is not calculable, because the number of participants with available values at this visit and treatment group is one.
  Cycle 8 Day 1: number analyzed (Participants) | 2 | 0 | 1 | 1
  Cycle 8 Day 1 | -2.10 (8.20) |  | -0.70 (NA) — The standard deviation is not calculable, because the number of participants with available values at this visit and treatment group is one. | -3.40 (NA) — The standard deviation is not calculable, because the number of participants with available values at this visit and treatment group is one.
  Cycle 9 Day 1: number analyzed (Participants) | 2 | 0 | 1 | 0
  Cycle 9 Day 1 | -2.10 (12.02) |  | -3.40 (NA) — The standard deviation is not calculable, because the number of participants with available values at this visit and treatment group is one. |
  Cycle 10 Day 1: number analyzed (Participants) | 2 | 0 | 1 | 0
  Cycle 10 Day 1 | 0.20 (7.78) |  | -1.10 (NA) — The standard deviation is not calculable, because the number of participants with available values at this visit and treatment group is one. |
  Cycle 11 Day 1: number analyzed (Participants) | 2 | 0 | 0 | 0
  Cycle 11 Day 1 | -0.75 (8.27) |  |  |
  Cycle 12 Day 1: number analyzed (Participants) | 2 | 0 | 1 | 0
  Cycle 12 Day 1 | 0.60 (7.21) |  | -2.30 (NA) — The standard deviation is not calculable, because the number of participants with available values at this visit and treatment group is one. |
  Cycle 13 Day 1: number analyzed (Participants) | 2 | 0 | 1 | 0
  Cycle 13 Day 1 | 1.00 (5.09) |  | -3.50 (NA) — The standard deviation is not calculable, because the number of participants with available values at this visit and treatment group is one. |
  Cycle 14 Day 1: number analyzed (Participants) | 1 | 0 | 1 | 0
  Cycle 14 Day 1 | 4.60 (NA) — The standard deviation is not calculable, because the number of participants with available values at this visit and treatment group is one. |  | -4.00 (NA) — The standard deviation is not calculable, because the number of participants with available values at this visit and treatment group is one. |
  Cycle 15 Day 1: number analyzed (Participants) | 1 | 0 | 1 | 0
  Cycle 15 Day 1 | 4.60 (NA) — The standard deviation is not calculable, because the number of participants with available values at this visit and treatment group is one. |  | 0.20 (NA) — The standard deviation is not calculable, because the number of participants with available values at this visit and treatment group is one. |
  Cycle 16 Day 1: number analyzed (Participants) | 0 | 0 | 1 | 0
  Cycle 16 Day 1 |  |  | -5.10 (NA) — The standard deviation is not calculable, because the number of participants with available values at this visit and treatment group is one. |
  Cycle 17 Day 1: number analyzed (Participants) | 0 | 0 | 1 | 0
  Cycle 17 Day 1 |  |  | -2.30 (NA) — The standard deviation is not calculable, because the number of participants with available values at this visit and treatment group is one. |
  EOT Visit: number analyzed (Participants) | 6 | 1 | 3 | 3
  EOT Visit | -1.67 (3.91) | 0.80 (NA) — The standard deviation is not calculable, because the number of participants with available values at this visit and treatment group is one. | 1.13 (4.14) | -4.67 (6.53)

8. Secondary Outcome: Response (Complete Response (CR) / CR According to iRECIST (iCR) / Partial Response (PR) / PR According to iRECIST (iPR)) and Stable Disease (SD) Duration - Arm A and Arm B
Description: Duration of stable disease is defined as the time from first diagnosis of response or stable disease (i.e., CR/iCR/PR/iPR/SD/iSD) to progression (i.e. progressive disease (PD), unconfirmed progressive disease according to iRECIST (iUPD), confirmed progressive disease (iCPD)) or death. Responding and stable patients without progression are censored at their last visit/study treatment administration. Patients who never respond or have a stable disease are excluded from this analysis.
Time Frame: Up to 36 months
Population: Only patients with response were analyzed. As in Arm B: Regimen 1: there was no patient with a response, the overall number of participants analyzed is 0.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Arm A: | Arm B: Regimen 1: | Arm B: Regimen 2: | Arm B: Regimen 3:
Number analyzed (Participants) | 2 | 0 | 3 | 4
days | 490.0 [462.0 to 518.0] |  | NA [43.0 to NA] — The median and upper confidence limit is not calculable because the number of participants with event is insufficient | 128.0 [43.0 to NA] — The upper confidence limit is not calculable because the number of participants with event is insufficient

9. Secondary Outcome: Plasma Concentration of Vilobelimab - Arm A and Arm B
Description: The plasma concentration of vilobelimab was assessed at different time points pre- and post-dose. The post-dose Cycle 1 Day 22 values correspond to Cmax and the pre-dose Cycle 1 Day 8, pre-dose Cycle 1 Day 22, pre-dose Cycle 2 Day 1 and per-dose Cycle 5 Day 1 values to Ctrough. In contrast to the time frame of the secondary efficacy outcome measures (3.-5., 7.-8), which were reported until EOS (up to 36 months), the time frames of ADAs (6.) and PK (9.) are measured (only) until first FU. Therefore, the time frame is different, i.e. 24 months of treatment until EOT + (approx.) 12 weeks/3 months until first FU up to 27 months.
Time Frame: Up to 27 months
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm A: | Arm B: Regimen 1: | Arm B: Regimen 2: | Arm B: Regimen 3:
Number analyzed (Participants) | 10 | 3 | 6 | 6
ng/mL
  Pre-dose Cycle 1 Day 8: number analyzed (Participants) | 9 | 3 | 6 | 6
  Pre-dose Cycle 1 Day 8 | 128404.2 (86.8) | 32488.5 (51.9) | 80525.0 (41.5) | 88749.9 (52.4)
  Pre-dose Cycle 1 Day 22 | 85088.6 (135.8) | 25312.8 (94.1) | 72792.5 (57.5) | 78248.6 (48.6)
  Post-dose Cycle 1 Day 22: number analyzed (Participants) | 9 | 3 | 6 | 6
  Post-dose Cycle 1 Day 22 | 514953.9 (43.5) | 208865.8 (27.6) | 261068.1 (96.7) | 210169.5 (66.1)
  Pre-dose Cycle 2 Day 1: number analyzed (Participants) | 7 | 1 | 4 | 6
  Pre-dose Cycle 2 Day 1 | 81260.1 (281.2) | 11124.0 (NA) — The geometric coefficient of variation is not calculable, because the number of participants with available values at this visit and treatment group is one | 48722.9 (106.9) | 80697.1 (104.1)
  Pre-dose Cycle 5 Day 1: number analyzed (Participants) | 2 | 0 | 1 | 2
  Pre-dose Cycle 5 Day 1 | 107989.9 (43.6) |  | 132497.0 (NA) — The geometric coefficient of variation is not calculable, because the number of participants with available values at this visit and treatment group is one | 41506.4 (65.9)

ADVERSE EVENTS:
Time Frame: Up to 36 months
Arm/Group | Arm A: | Arm B Regimen 1: | Arm B Regimen 2: | Arm B Regimen 3:
All-Cause Mortality (participants affected / at risk) | 7/10 | 2/3 | 4/6 | 1/6
Serious Adverse Events (participants affected / at risk) | 7/10 | 2/3 | 2/6 | 1/6
Other Adverse Events (participants affected / at risk) | 9/10 | 3/3 | 5/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: (N=10) | Arm B Regimen 1: (N=3) | Arm B Regimen 2: (N=6) | Arm B Regimen 3: (N=6)
General physical health deterioration (General disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac Failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amyloidosis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: (N=10) | Arm B Regimen 1: (N=3) | Arm B Regimen 2: (N=6) | Arm B Regimen 3: (N=6)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Asthenia (General disorders) | 2 (2) | 0 (0) | 1 (2) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Infusion site paraesthesia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dental discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral hyperkeratosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection pseudomonas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Dementia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intraocular pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thyroxine free increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin discharge (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoradionecrosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Traumatic haematome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Skin neoplasm bleeding (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphorrhoea (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scalp haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was prematurely terminated due to a strategic decision by the sponsor. Therefore, the total number of participants enrolled is smaller than planned (actually enrolled and treated: 25, planned: 70).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-12): https://cdn.clinicaltrials.gov/large-docs/35/NCT04812535/Prot_SAP_000.pdf